CLINICAL TRIAL: NCT05197725
Title: Face Masks to Reduce Symptomatic and Asymptomatic SARS-CoV-2 Infections in Bangladesh
Brief Title: Face Masks to Reduce SARS-CoV-2 Infections (COVID-19) in Bangladesh
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to get Study supplies in time
Sponsor: Yale University (Other)
Collaborators: Stanford University (Other); University of California, Berkeley (Other); Innovations for Poverty Action (Other); North South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2000028482_asymp; INV-037905 (Other Grant/Funding Number: Gates Foundation)
Record Dates: First submitted 2022-01-14; First posted 2022-01-19 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Covid19
Keywords: Masks; Transmission; Bangladesh; Behavioral psychology
MeSH Terms: conditions — COVID-19 | interventions — Masks

STUDY DESIGN:
Intervention Model Description: This is a randomized controlled trial with an equal number of intervention and control villages enrolled each day.
Who Masked: Investigator
Masking Description: The intervention involves wearing a face mask so participants will know if they are in the intervention group. The investigators will be blinded as to intervention assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mask intervention (Experimental): Communities randomized to the intervention arm will be given masks and behavior change communication to motivate proper mask use. Every adult in communities randomized to the intervention arm will be encouraged to wear a mask when outside their housing compound and around other people. In arms randomized to school promotion, secondary school children will also be encouraged to wear masks both inside and outside of school.
  Interventions: Device: Face mask; Behavioral: Face mask awareness; Behavioral: Face mask promotion through community values or individual information
- Control (No Intervention): Control individuals will receive no masks or behavior change communication.

INTERVENTIONS:
Device: Face mask — Individuals in intervention communities will be given surgical or KF94 face masks.
  Arms: Mask intervention
Behavioral: Face mask awareness — Intervention individuals will be told about the importance of wearing face masks that cover the nose, mouth, and chin. Mask by mask promoters and community and religious leaders will encourage mask wearing.
  Arms: Mask intervention
Behavioral: Face mask promotion through community values or individual information — In intervention communities randomized to mask promotion through community values, promotional discussions and media will focus on encouraging groups of people to wear masks as a reflection of their values.
  In intervention communities randomized to mask promotion through individual information, promotional discussions and media will target individuals and focus on the instrumental value of wearing masks (preventing the inhalation of viral particles)
  Arms: Mask intervention

SUMMARY:
The primary goal of the village-level intervention is to assess whether mask-wearing reduces community-level asymptomatic and symptomatic SARS-CoV-2 infections, assessed via PCR testing. The study also examines if community-based activation through values or individual activation through information results in higher mask-wearing.

DETAILED DESCRIPTION:
Detailed Description:

This study intends to answer the following research questions:

Can mask distribution and mask promotion at homes, mosques, markets and other public areas successfully change community mask-wearing norms to increase mask-wearing, even years into a pandemic?

Can community mask-wearing reduce SARS-CoV-2 infections (both symptomatic and asymptomatic)?

Is increased prevalence of community-level mask-wearing associated with decreased physical distancing?

To answer these questions, the investigators will conduct a cluster randomized trial which randomizes the proposed intervention at the village level in Bangladesh. Control communities will receive no intervention and treatment communities will receive an extensive intervention combining several elements. Study staff will distribute free face masks through door-to-door visits and at markets and mosques. In some communities groups of people will be encouraged to wear masks by appealing to their shared values and in other communities individuals will be encouraged to wear masks by discussing the biological value of masks (cross-randomized among intervention communities). Mask promoters in the community and at markets in treated villages will remind people about the importance of wearing masks and distribute additional masks. Markets will have signs that masks need to be worn to enter the market. Religious leaders will encourage mask use at religious services. The project will enroll 1200 communities, stratified in geographically proximate groups of 10; half will be randomized to receive the intervention.

Communities will be surveilled through direct observation at 0, 2, and 4 weeks to assess mask-wearing. The investigators will assess symptomatic and asymptomatic SARS-CoV-2 by conducting household visits every 6-10 days to ask about symptoms of COVID-19 and collecting nasal swabs to test by PCR for the presence of SARS-CoV-2. End line is planned for 4 weeks after the intervention begins, but may be shifted according to seroprevalence trends.

ELIGIBILITY:
Inclusion Criteria:

* Live in selected village

Exclusion Criteria:

* None

Min Age: 12 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-02-04 (Estimated); Primary Completion 2023-03-30 (Estimated); Study Completion 2023-05-30 (Estimated)

PRIMARY OUTCOMES:
Asymptomatic and asymptomatic SARS-CoV-2 infection | approximately weekly for 4 weeks; may be lengthened if the intervention is extended due to low than estimated seroprevalence at the start of the intervention
  Asymptomatic and asymptomatic SARS-CoV-2 infection, assessed using PCR testing every 6-10 days after baseline, among individuals regardless of whether they report symptoms of COVID-19

SECONDARY OUTCOMES:
Observed prevalence of mask-wearing | Intervention weeks 0, 2, and 4; end line and midline timepoints may be adjusted if the intervention is extended due to low than estimated seroprevalence at the start of the intervention.
  Percent of people observed in public places wearing a mask over their mouth and nose compared to wearing a mask or face covering that does not cover the mouth and nose or not wearing any mask or face covering. The investigators will include sub-group analyses by age group, gender, and location
Respiratory infection prevalence | approximately weekly for 4 weeks; may be lengthened if the intervention is extended due to low than estimated seroprevalence at the start of the intervention
  Prevalence of self-reported symptoms of COVID-19, including fever, cough, sore throat, shortness of breath, difficulty breathing, nasal congestion, and runny nose.
Physical distancing | Intervention weeks 0, 2, and 4; end line and midline timepoints may be adjusted if the intervention is extended due to low than estimated seroprevalence at the start of the intervention.
  Prevalence of physical distancing among observed individuals wearing or not wearing a mask

CONTACTS AND LOCATIONS:
Locations (1):
- Innovations for Poverty Action, Dhaka, Bangladesh

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to share individual participant data with other researchers

DOCUMENTS (2):
  • Study Protocol (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/25/NCT05197725/Prot_001.pdf
  • Informed Consent Form (2022-01-06): https://cdn.clinicaltrials.gov/large-docs/25/NCT05197725/ICF_000.pdf